CLINICAL TRIAL: NCT01269203
Title: A Phase II Randomized Study of the Efficacy of Curcumin for Reducing Symptoms During Maintenance Therapy in Multiple Myeloma Patients
Brief Title: Efficacy of NF-kB Inhibition for Reducing Symptoms During Maintenance Therapy in Multiple Myeloma Patients
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 2010-0457
Record Dates: First submitted 2010-12-30; First posted 2011-01-04 (Estimated); Last update posted 2012-09-07 (Estimated); Status verified 2012-09

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma; MM; maintenance therapy; lenalidomide; bone marrow transplantation; auto-HSCT; Autologous Hematopoietic Stem Cell Transplantation; NF-kB inhibition; reducing symptoms; maintenance chemotherapy; inflammatory cytokines; nuclear factor kappa B; NF-kB; interleukin; IL-6; tumor necrosis factor; TNF-a; NF-kB activation levels
MeSH Terms: conditions — Multiple Myeloma | interventions — Curcumin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Curcumin (Active Comparator): 1000 mg/day Curcumin + 5 -15 mg/day Lenalidomide
  Interventions: Drug: Curcumin
- Placebo (Placebo Comparator): Placebo daily + 5 -15 mg/day Lenalidomide
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Curcumin — 1000 mg per day
  Arms: Curcumin
Other: Placebo — Administered daily same as Curcumin.
  Arms: Placebo

SUMMARY:
The goal of this clinical research study is to learn if curcumin can reduce the symptoms reported by patients with multiple myeloma (MM) who receive treatment with lenalidomide.

DETAILED DESCRIPTION:
Curcumin is the active ingredient in the spice turmeric. It may interfere with the production of cytokines (which cause inflammation), which may help reduce multiple symptoms.

A placebo is not a drug. It looks like the study drug but is not designed to treat any disease or illness. It is designed to be compared with a study drug to learn if the study drug has any real effect.

Study Groups:

If you agree to take part in this study, you will be randomly assigned (as in the flip of a coin) to 1 of 2 groups. Group 1 will take curcumin. Group 2 will take a placebo. You will have an equal chance of being assigned to each group. No matter which group you are in, you will be given standard care by your treating doctor.

Neither you nor the study staff will know if you are receiving the study drug or the placebo. However, if needed for your safety, the study staff will be able to find out what you are receiving.

Study Drug Administration:

You will take curcumin/placebo 2 times every day about 12 hours apart. You will begin taking curcumin/placebo when you begin maintenance therapy with lenalidomide.

You will be given a pamphlet with more information about how to take the curcumin/placebo.

You must bring the study capsules you have not yet taken to the clinic every study visit.

Every 4 weeks is called a study cycle.

Study Visits:

Before you begin treatment with lenalidomide and curcumin/placebo:

* You will be taught how to use the automated symptom assessment telephone program.
* You will complete 4 questionnaires about pain and other symptoms, and your quality of life. In addition, some personal information (such as your name, address, race, and smoking history) will be collected. Completing the questionnaires will take about 20 minutes.
* You will be asked about any drugs you may be taking.
* You will be asked how well you are able to perform the normal activities of daily living (performance status).

Telephone System Calls for Symptom Monitoring:

A telephone system will call you once a week at a time convenient to you. Using the numeric key pad on your telephone, you will rate your symptoms and how they interfere with your daily activities. Each phone call will take about 5 minutes to complete. You will be given a brochure explaining the steps to complete the symptom questionnaire and a telephone number to call if you have questions or problems with the telephone system.

At the start of Cycle 4 and at the End of Study Visit:

-You will complete 3 questionnaires about your pain and other symptoms and your quality of life. The questionnaires will take about 20 minutes to complete. If for some reason, you are unable to complete the questionnaire through the automated symptom assessment telephone program, you may be able to complete it with the research staff, either by phone or during a routine clinic visit.

Research staff will talk to you during your regularly scheduled visits for each cycle of treatment with lenalidomide. You will be asked about side effects you may be having and drugs you are taking.

Length of Study:

You will take curcumin/placebo for 6 months. You will remain on the study for about 6-7 months (depending on how your clinic visits are scheduled). You will be taken off study if you have intolerable side effects or the disease gets worse.

This is an investigational study. Curcumin is not FDA approved. At this time, curcumin is only being used in research.

Up to 70 participants will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Must have a histologically confirmed diagnosis of multiple myeloma.
2. Must be >/= 18 years of age.
3. Must have a performance status (ECOG PS) of 0-2.
4. Must be qualified and have signed consent to receive lenalidomide for maintenance therapy for MM.
5. Must have signed informed consent indicating that they are aware of the investigational nature of the study, and are aware that participation is voluntary.
6. Must also agree to refrain from use of self prescribed curcumin during the course of the study.
7. Must have negative pregnancy test before signing consent for MM therapy.

Exclusion Criteria:

1. Unable to understand the symptom assessment or not willing to participate in the study.
2. Treatment for other carcinomas within the last 5 years, except for cured non-melanoma skin and treated in-situ cervical cancer.
3. Uncontrolled intercurrent illness including, but not limited to, ongoing or requiring IV antibiotics, cardiac disease (NYHA class III or IV heart failure), unstable angina pectoris, unstable cardiac arrhythmia or tachycardia, or psychiatric illness/ social situations that would limit compliance with the study requirements are excluded.
4. Concurrent use of coumadin other than low dose (1 mg) coumadin used for line patency.
5. Concurrent use of cimetidine, allopurinol, or aluminium hydroxide and magnesium hydroxide-containing antacids such as Maalox.
6. Sorivudine and brivudine use within 4 weeks of the start of study treatment.
7. Gastric or duodenal ulcers, or gastric hyperacidity disorders.
8. Currently receiving anticoagulants (heparin) or antiplatelets (clopidogrel, ticlopidine, aspirin/dipyridamole)
9. INR > 1.5 (upper limit of normal = 1.5).
10. History of deep vein thrombosis.
11. Received allogeneic transplant.
12. Allergy to turmeric, Curcumin, or yellow dye.
13. Bowel or bile duct obstruction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-10; Primary Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
AUC from 3 months Post-Transplantation to 9 months Post-Transplantation | Assessments within +/-3 days of 4 week cycle start date for 6 cycles.
  Daily area under the curve (AUC) where AUC is based on average of 5 most severe symptoms (pain, fatigue, bone aches, numbness, disturbed sleep) being experienced by MM patients as measured by MDASI-MM, a multiple-symptom measure of cancer-related symptoms rate severity of physical, affective, and cognitive symptoms on 0-10 numeric scales, ranging from 0 "not present" to 10 "as bad as you can imagine."

CONTACTS AND LOCATIONS:
Overall Officials: Robert Orlowski, MD, PhD, Study Chair — UT MD Anderson Cancer Center

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org